CLINICAL TRIAL: NCT04823338
Title: Conectar Jugando Online: Effectiveness of an Online Modern Board Game-based Cognitive Training to Improve Executive Function in School-age Children by a Randomized Controlled Trial
Brief Title: Conectar Jugando Online: Board Games to Improve Executive Function in School-age Children (CJ-Online)
Acronym: CJ-Online
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brain In Game scientific-technical service (Other)
Collaborators: Atención, Familia, Infancia, Mayores (AFIM21) (Unknown); Mercurio Distribuciones (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NCT2021CJ
Record Dates: First submitted 2021-03-23; First posted 2021-03-30 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Cognitive Change; Child Development
Keywords: executive function; modern board and card games; cognitive training; school-age children

STUDY DESIGN:
Intervention Model Description: Interventional (Clinical trial)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conectar Jugando Online Program (Experimental): The program consisted of 12 one-hour intervention sessions. The sessions were biweekly with a total duration of 6 weeks. The modern board and card games used in the program were Bee Alert (Knizia, 2012), Monster Match (Gruhl & Weir, 2018), Sherlock Express (Kermarrec, 2019), Streams (Itsubaki, 2011) and Blurble (Bernard, 2013). The play sessions were carried out in groups of between 2 and 4 boys and girls of similar ages (same school stage) formed according to the availability of the participants. In the sessions, the physical games were projected on the videoconference tool by the researcher and the participating boys and girls carried out their actions using their voice and the platform tools. The program was gamified though a narrative about a space travel to different planets in discovering new games and get different mission badges and super team badges in their logbook.
  Interventions: Behavioral: Conectar Jugando Online Program
- Wait-list group (No Intervention): Wait-list

INTERVENTIONS:
Behavioral: Conectar Jugando Online Program — Online play sessions with modern board and card games guided by the study researchers
  Other Names: Modern board and card games
  Arms: Conectar Jugando Online Program

SUMMARY:
Good development of executive functions at school has been related to a better adaptation of children in different areas of their daily life and, especially, with adequate academic performance. Taking into account the importance of play in childhood, some interventions aimed at training these cognitive processes have been based on the use of playful elements, such as modern board games. Although it is still an unexplored field of research, some studies with older elementary school children and with ADHD children have found significant improvements in executive functions after training that had the board game as a key intervention element. However, we still do not have studies that have explored the possible cognitive benefits of its use throughout the primary stage with the general population. For this reason, the main objective of this study is to test the effectiveness of a cognitive training program based on modern board games in primary education children (6 to 12 years old).

DETAILED DESCRIPTION:
As hypotheses, it is established that: i) the experimental group will present a significantly greater improvement in the neuropsychological tasks that measure executive functions and associated cognitive processes compared to the passive control group after the intervention; ii) the experimental group will present a significantly greater improvement in the tests evaluated by their parents after the intervention compared to the passive control group. All hypotheses will be controlled for age, estimate of IQ and socioeconomic status, as well as previous experience in board games and other cognitive activities.

ELIGIBILITY:
Inclusion Criteria:

* be enrolled in a public, private or subsidized ordinary educational center
* provide informed consent from both parents and the participant's agreement to participate in the study

Exclusion Criteria:

* comprehension difficulties due to language reasons
* sensory difficulties that make it impossible to carry out the program activities
* not having the necessary equipment to monitor the sessions online

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-06-16 (Actual)

PRIMARY OUTCOMES:
Change in verbal updating from baseline to post intervention | Baseline and post intervention (after 6 weeks)
  Verbal keep track task (Tamnes et al., 2010)
Change in visuospatial updating from baseline to post intervention | Baseline and post intervention (after 6 weeks)
  Visuospatial keep track task (Tamnes et al., 2010)
Change in inhibition from baseline to post intervention | Baseline and post intervention (after 6 weeks)
  5 digits test (Sedó, 2004)
Change in cognitive flexibility from baseline to post intervention | Baseline and post intervention (after 6 weeks)
  5 digits test (Sedó, 2004)
Change in reasoning from baseline to post intervention | Baseline and post intervention (after 6 weeks)
  TONI-4 (Ruíz-Fernández, 2019)
Change in verbal fluency from baseline to post intervention | Baseline and post intervention (after 6 weeks)
  Phonological and semantic fluency (letter M and animals, ENFEN, Portellano & Martínez-Arias, R. Zumárraga, 2009)

SECONDARY OUTCOMES:
Change in behavioral executive functions from baseline to post intervention | Baseline and post intervention (after 6 weeks)
  ATENTO (Luque & Sánchez-Sánchez, 2019)
Change in emotional and behavioral problems from baseline to post intervention | Baseline and post intervention (after 6 weeks)
  SENA (Sistema de Evaluación de Niños y Adolescentes, Fernández-Pinto, L Santamaría, Sánchez-Sánchez, F Carrasco, & Del Barrio, 2015)

OTHER OUTCOMES:
Time spent on less-structured activities | Baseline
  adapted from "Parent Survey of Typical Child Time Spent in Less-structured Activities" (Barker et al., 2014) In this survey, parents are asked (with the help of their children) about the time their children dedicate to less-structured and recreational activities using a using a 7-point scale (from lowest to highest frequency). High scores on each item mean a higher frequency in that activity. The sum of all the scores on each item (where 1= 'Never' and 7 = 'Daily') results in a typical less-structured activity score.
Player satisfaction | During the intervention
  Visual analogue scale created ad hoc
  The scale consists of two questions:
  * Degree of satisfaction in reference to the play session
  * Degree of satisfaction in reference to the modern board and card games used in the play session Participants respond using a 5-option scale consisting of 5 stars (1 star = Not at all satisfied; 5 = Very satisfied)
Sociodemographic data (age, sex, school year and socioeconomic status) | Baseline
  Hollingshead Index (Hollingshead, 1975)
Parent Play Beliefs | Baseline and post intervention (after 6 weeks)
  "The Parent Play Beliefs Scale (PPBS)" (Fogle & Mendez, 2006) It consists of 30 items with 5 response options ranging from 1 (Disagree) to 5 (Strongly agree). Two subscales have been considered: a) Play support; b) Acedemic focus.
  The Play Support subscale refers to parents' positive beliefs about the relevance of play for children's development and about their participation in play with children. High scores on this subscale indicate that parents enjoy play, prioritize play, and view it as a means of teaching.
  The Academic focus subscale is made up of elements about the parents' emphasis on academic skills and the belief that play can promote their development. The Academic focus subscale is made up of elements about the parents' emphasis on academic skills and the belief that play can promote their development. High scores on this subscale would indicate that parents see the academic role of play as important.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Education, Psychology and Social Work; University of Lleida, Lleida, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Benzing V, Schmidt M, Jager K, Egger F, Conzelmann A, Roebers CM. A classroom intervention to improve executive functions in late primary school children: Too 'old' for improvements? Br J Educ Psychol. 2019 Jun;89(2):225-238. doi: 10.1111/bjep.12232. Epub 2018 Jun 26. PMID 29947142
- [Background] Diamond A. Executive functions. Annu Rev Psychol. 2013;64:135-68. doi: 10.1146/annurev-psych-113011-143750. Epub 2012 Sep 27. PMID 23020641
- [Background] Estrada-Plana V, Esquerda M, Mangues R, March-Llanes J, Moya-Higueras J. A Pilot Study of the Efficacy of a Cognitive Training Based on Board Games in Children with Attention-Deficit/Hyperactivity Disorder: A Randomized Controlled Trial. Games Health J. 2019 Aug;8(4):265-274. doi: 10.1089/g4h.2018.0051. Epub 2019 Jan 17. PMID 30653355
- [Background] Fadhli, M., Brick, B., Setyosari, P., Ulfa, S., & Kuswandi, D. (2020). A Meta-Analysis of Selected Studies on the Effectiveness of Gamification Method for Children. International Journal of Instruction, 13(1), 845-854. https://doi.org/10.29333/iji.2020.13154a